CLINICAL TRIAL: NCT00930111
Title: Inpatient Attending Physician Rotation Duration Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamela Gonzalez Sr Director Clinical Research Office (Other Government)
Responsible Party: Sponsor-Investigator, Pamela Gonzalez Sr Director Clinical Research Office, Dir Clinical Research, Cook County Health
Organization: Cook County Health (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 09-063 Cooker 533
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Inpatient Attending Physician Staffing Model
Keywords: inpatient; hospitalists; residency; job satisfaction; burnout, professional; professional practice; medical education
MeSH Terms: conditions — Burnout, Professional | interventions — Rotation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 weeks (Active Comparator): Attending physicians are physician-of-records for traditional inpatient ward team (housestaff and medical students) for 2 weeks.
  Interventions: Other: 2-week rotation
- 4 weeks (Placebo Comparator): Attending physicians are physician-of-records for traditional inpatient ward team (housestaff and medical students) for 4 weeks.
  Interventions: Other: 4-week rotation

INTERVENTIONS:
Other: 2-week rotation — Attending physician is assigned to a 2-week rotation.
  Arms: 2 weeks
Other: 4-week rotation — Attending physician is assigned to a 4-week rotation.
  Arms: 4 weeks

SUMMARY:
The investigators are testing the effects of a change in teaching attending physicians' rotations (from 4- to 2-week blocks) on patient outcomes (unplanned urgent visits to the health care system, inpatient mortality, and length-of-stay), the educational experiences of residents and medical students and on the quality of the professional lives of the attending physicians.

DETAILED DESCRIPTION:
Design, Setting, and Participants Cluster randomized crossover noninferiority trial, with attending physicians as the unit of crossover randomization and 4-week rotations as the active control, conducted in a US university-affiliated teaching hospital in academic year 2009. Participants were 62 attending physicians who staffed at least 6 weeks of inpatient service, the 8892 unique patients whom they discharged, and the 147 house staff and 229 medical students who evaluated their performance.

Intervention Assignment to random sequences of 2- and 4-week rotations.

Main Outcome Measures Primary outcome was 30-day unplanned revisits (visits to the hospital's emergency department or urgent ambulatory clinic, unplanned readmissions, and direct transfers from neighboring hospitals) for patients discharged from 2- vs 4-week within-attending-physician rotations. Noninferiority margin was a 2% increase (odds ratio [OR] of 1.13) in 30-day unplanned patient revisits. Secondary outcomes were length of stay; trainee evaluations of attending physicians; and attending physician reports of burnout, stress, and workplace control.

ELIGIBILITY:
Inclusion Criteria:

* Attending physician on inpatient general medicine wards of Stroger Hospital, Chicago, IL

Exclusion Criteria:

* Scheduled for less than 6 weeks during the 2009 academic year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-06; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Patients' unplanned urgent visits to the health care system. | 30 days after discharge
  Number pf non-scheduled patient encounters documented in the EHR

SECONDARY OUTCOMES:
Resident physicians' evaluation of attending physicians' performance. | During 14 or 28 day rotations
  Self administered performance electronic evaluations - validated tool
Medical students' evaluations of attending physicians' performance. | During 14 or 28 day rotations
  Self administered performance electronic evaluations
Urgent visits to health care system among attending physicians' outpatient panel (if attending physician has an outpatient panel) | During and 14 to 28 days after provider's rotation
  Number pf non-scheduled patient encounters documented in the EHR
Attending physicians' work-life balance, perceived stress, and perceived burn-out. | During 14 to 28 day rotations
  Self administered confidential Burnout assessment survey based on Conceptual Model of Burnout, Perceived Stress Scale & Maslach Burnout Inventory Human ServiceSurvey and a single item measure from the Notional Job Burnout Survey.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lucas, MD, Principal Investigator — Cook County Health
Locations (1):
- Stroger Hospital of Cook County, Chicago, Illinois, United States

REFERENCES:
- [Derived] Lucas BP, Trick WE, Evans AT, Mba B, Smith J, Das K, Clarke P, Varkey A, Mathew S, Weinstein RA. Effects of 2- vs 4-week attending physician inpatient rotations on unplanned patient revisits, evaluations by trainees, and attending physician burnout: a randomized trial. JAMA. 2012 Dec 5;308(21):2199-207. doi: 10.1001/jama.2012.36522. PMID 23212497